CLINICAL TRIAL: NCT04029051
Title: Focus Thoracic Ultrasound for Dyspnea Diagnosis in Elderly Patient in the ED: Prospective Observational Study
Brief Title: Focus Thoracic Ultrasound for Dyspnea Diagnosis in Elderly Patient in the Emergency Department
Acronym: echoelderly
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-036
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Dyspnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Focus thoracic ultrasound for dyspnea diagnosis — Focus thoracic ultrasound is composed by an advanced cardiac ultrasound with Doppler measures and a lung ultrasound.

SUMMARY:
Brief Summary: The aim of this study is to analyze in elderly patients with undifferentiated dyspnea, the concordance of diagnosis before and after a focus thoracic ultrasound in comparison with the reference one established by an adjudication committee

DETAILED DESCRIPTION:
Dyspnea is associated with a variety of etiology whose diagnosis is challenging especially in elderly patients with unconventional symptoms. Focus thoracic ultrasound is composed by an advanced cardiac ultrasound with Doppler measures and a lung ultrasound. It has already demonstrated its ability to reduce diagnosis uncertainty in emergency patients with dyspnea. However, adequacy of diagnosis before and after thoracic ultrasound has not been investigated in such patients.

In this population, after clinical examination and use of any resource deemed necessary, the physician states its hypothesis in closed list. An emergency physician then realizes a thoracic ultrasound exam. An adjudication committee with all the patient's file will state the reference hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Acute onset dyspnea in patient over 74 years old consulting at the emergency department

Exclusion Criteria:

* Need for ICU
* Need for a mechanical ventilation
* Less than 24 hours hospital stay
* Inability to consent

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patient consulting in the emergency department for acute onset dyspnea
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
main objective | 3 years
  Concordance between initial diagnosis after standard care, after thoracic ultrasound in comparison with the reference stated by the adjudication committee

SECONDARY OUTCOMES:
Frequency | 3 years
  Frequency of each diagnosis in elderly patients consulting in the emergency department
mortality | 3 years
  Assessing hospital mortality in elderly patients consulting at the emergency department

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Carvalho H, Javaudin F, Le Bastard Q, Boureau AS, Montassier E, Le Conte P. Effect of chest ultrasound on diagnostic workup in elderly patients with acute respiratory failure in the emergency department: a prospective study. Eur J Emerg Med. 2021 Jan 1;28(1):29-33. doi: 10.1097/MEJ.0000000000000732. PMID 32568788